CLINICAL TRIAL: NCT04162925
Title: Cancer Screening Utilization Rates and Cancer Screening Perspectives of Hospitalized Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: State of Maryland (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00049608; IO90059879 (Other Grant/Funding Number: State of Maryland)
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Cancer Screening

STUDY DESIGN:
Intervention Model Description: Cancer screening utilization rates and cancer screening perspective of hospitalized women on internal medicine service
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer screening cohort (Experimental): All women in this study to be evaluated for cancer screening utilization rates (breast, colon and oral cancers) and cancer screening perspectives of these hospitalized women.
  The intervention will be a cancer screening education.
  Interventions: Behavioral: Cancer screening education for breast, colon and oral cancers

INTERVENTIONS:
Behavioral: Cancer screening education for breast, colon and oral cancers — Bedside education one-on-one by showing screening video and handouts at the end of educational session for breast, colon and oral cancer. Patient who are agreeable to oral cancer screen during hospitalization perform oral cancer screening

SUMMARY:
Breast and colon cancers are commonly diagnosed cancers among women after skin cancer in Maryland. Patients' preferences for cancer screening are known to significantly influence utilization, and thus impact health outcomes. In a recent study the investigators conducted at Johns Hopkins Bayview Medical Center, the investigators observed that among women age 50-75 years admitted to general medicine services over 4-month period, 40% were non-adherent to breast cancer screening (overdue) despite being insured.

Therefore, the investigators propose to establish a cohort of hospitalized women to help the investigators develop successful interventions for enhancing breast cancer screening utilization in this group. In following a cohort prospectively, the investigators intend to both reaffirm the results from the investigators' previous study and determine whether the patterns of mammographic screening improve over time as a result of the investigators' interventions. Among non-adherent (overdue) women, the investigators will educate and encourage these women to undergo outpatient screening mammography.

To more comprehensively assess the preventive health in this cohort, the investigators will assess the cohort's adherence to colon cancer screening recommendation and barriers to colon cancer screening.

In addition the investigators will also like to encourage the hospitalists and house staff taking care of these patients to perform oral cancer screen among women who smoke (non-adherent to breast cancer screening) Finally the investigators will also like to ask the perspective of cancer screening among these women.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 50 to 75 years admitted to medicine service at Johns Hopkins Bayview Medical Center
* cancer free at baseline (excluding skin cancers)
* willing to participate voluntarily

Exclusion Criteria:

* history of breast cancer or mastectomy
* history of other cancers (except skin) or serious comorbidities making life expectancy <10 years
* pregnancy
* dementia
* chronic disability (unable to stand or nursing home resident)
* current admission because of acute coronary event (heart attack) or stroke or pulmonary embolism
* chronic kidney disease on hemodialysis
* history of BRCA1 or BRCA2 gene mutation
* current admission for cellulitis or abscess of breast

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — hospitalized women between ages of 50-75 who will be cancer free at the time of enrollment (except for skin cancer)
Enrollment: 700 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of women non-adherent to breast cancer screening in this group | 3 years
  Proportion of women non-adherent to breast cancer screening will be assessed in these hospitalized women.
Prevalence of breast cancer screening post intervention in this group | 3 years
  Prevalence of breast cancer screening post intervention will be assessed in these hospitalized women.
Proportion of hospitalized women non-adherent to colon cancer screening | 3 years
  Proportion of hospitalized women non-adherent to colon cancer screening will be assessed in these hospitalized women.
Perspective of hospitalized women about colon cancer screening as assessed by multiple choice questions | 3 years
  survey of hospitalized women using multiple choice 21 questions
Perspective of hospitalized women about colon cancer screening as assessed by likert scale 21 questions | 3 years
  survey of hospitalized women using likert scale 21 questions
Proportion of women non-adherent to oral cancer screening | 3 years
  Proportion of women non-adherent to oral cancer screening will be assessed in these hospitalized women.
Number of women agreeable to inpatient oral cancer screening exam | 3 years
  oral cavity screening exam consisting of mouth and neck examination by hospital providers
Perspective of hospitalized women in general about their preference for cancers screening as assessed by multiple choice questions | 3 years
  a survey consisting of 55 multiple choice questions
Perspective of hospitalized women in general about their preference for cancers screening as assessed by likert scale | 3 years
  a survey with a likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Khaliq, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olayinka O, Gnanaraj J, Khaliq W. Hospitalized Women's Willingness to Pay for Inpatient Screening Colonoscopy. Womens Health Rep (New Rochelle). 2022 Sep 13;3(1):768-773. doi: 10.1089/whr.2022.0014. eCollection 2022. PMID 36185070